CLINICAL TRIAL: NCT04797338
Title: Luteal Phase Support Using Gonadotropin Releasing Hormone Agonist (GnRHa) Versus Estrogen and Progesterone Supplementation in High Responders Following GnRHa Triggering - A Prospective Randomized Controlled Trial
Brief Title: Gonadotropin Releasing Hormone Agonist (GnRHa) Versus Estrogen and Progesterone for Luteal Support in High Responders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, principal investigator, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0245-17-ASF
Record Dates: First submitted 2021-03-03; First posted 2021-03-15 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy Early; Miscarriage; Ovarian Hyperstimulation Syndrome
MeSH Terms: conditions — Abortion, Spontaneous; Ovarian Hyperstimulation Syndrome | interventions — Nafarelin; estradiol, estriol drug combination; Estradiol; Utrogestan; Progesterone; 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Intervention Model Description: A randomization list will be generated by a computer by 1:1 ratio. Sealed envelopes containing treatment allocation instructions will be attached to the consent forms.
  At the day of triggering for final oocyte maturation, patients will sign an informed consent and will be allocated to one of the study arms according to the instructions in the envelop attached to the consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GnRHa treatment based luteal support (Active Comparator): Patients will initiate intranasal treatment with Nafarelin inhaler: 200 micrograms twice daily (a total of 400 micrograms/d; Synarel, Pfizer) on the evening after oocyte retrieval which will be continued up to the bHCG blood test, 12 days post embryo transfer. In cases with positive serum hCG results, the treatment will be stopped.
  Interventions: Drug: Synarel, 0.2 Mg/Inh Nasal Spray
- Estrogen and progesterone supplementation (Active Comparator): Patients will start treatment with a combination of oral estrogen (Estrofem or Progynova 4 mg twice daily), vaginal progesterone (vaginal Utrogestan 200mg or Endometrin 100 mg three times daily) and intramuscular injection of progesterone retard 250 mg once every five days. The treatment will start at the day of the oocyte retrieval up to the bHCG blood test, 12 days post embryo transfer. In cases with positive serum hCG results, the treatment will be continued up to 9+0 weeks of pregnancy.
  Interventions: Drug: Estrofem; Drug: Utrogestan; Drug: Hydroxyprogesterone Caproate

INTERVENTIONS:
Drug: Synarel, 0.2 Mg/Inh Nasal Spray — Intranasal treatment with Nafarelin inhaler: 200 micrograms twice daily (a total of 400 micrograms/d; Synarel, Pfizer) on the evening after oocyte retrieval, which will be continued up to the bHCG blood test, 12 days post embryo transfer. In cases with positive serum bHCG results, the treatment will be stopped.
  Other Names: Nafarelin
  Arms: GnRHa treatment based luteal support
Drug: Estrofem — A combination of oral estrogen (Estrofem or Progynova 4 mg twice daily), vaginal progesterone (vaginal Utrogestan 200mg or Endometrin 100 mg three times daily) and intramuscular injection of Hydroxyprogesterone Caproate 250 mg once every five days. The treatment will start at the day of the oocyte retrieval up to the bHCG blood test, 12 days post embryo transfer. In cases with positive serum bHCG results, the treatment will be continued up to 9+0 weeks of pregnancy.
  Other Names: Progynova
  Arms: Estrogen and progesterone supplementation
Drug: Utrogestan — A combination of oral estrogen (Estrofem or Progynova 4 mg twice daily), vaginal progesterone (vaginal Utrogestan 200mg or Endometrin 100 mg three times daily) and intramuscular injection of Hydroxyprogesterone Caproate 250 mg once every five days. The treatment will start at the day of the oocyte retrieval up to the bHCG blood test, 12 days post embryo transfer. In cases with positive serum bHCG results, the treatment will be continued up to 9+0 weeks of pregnancy.
  Other Names: Endometrin
  Arms: Estrogen and progesterone supplementation
Drug: Hydroxyprogesterone Caproate — A combination of oral estrogen (Estrofem or Progynova 4 mg twice daily), vaginal progesterone (vaginal Utrogestan 200mg or Endometrin 100 mg three times daily) and intramuscular injection of Hydroxyprogesterone Caproate 250 mg once every five days. The treatment will start at the day of the oocyte retrieval up to the bHCG blood test, 12 days post embryo transfer. In cases with positive serum bHCG results, the treatment will be continued up to 9+0 weeks of pregnancy.
  Other Names: Proluton Depot
  Arms: Estrogen and progesterone supplementation

SUMMARY:
Gonadotropin Releasing Hormone agonist (GnRHa) triggering is used as an alternative to human chorionic gonadotropin (hCG) in GnRH antagonist protocol to eliminate the risk of ovarian hyperstimulation syndrome (OHSS). However, its main disadvantage is a significantly lower pregnancy rate, hypothesized to result from a process called "luteolysis" (demise of the corpora lutea). In order to preserve a high pregnancy rates, several luteal support regimens were investigated, including an intensive estrogen and progesterone supplementation and a daily GnRHa treatment. However, no study, so far, compared the efficacy of these two regimens. Our aim is to compare the efficacy of GnRHa versus estrogen and progesterone supplementation for luteal phase support in high responders following GnRHa triggering.

DETAILED DESCRIPTION:
The administration of human chorionic gonadotropin (hCG) for final oocyte maturation is an accepted practice in in vitro fertilization (IVF) treatments. However, in high-responder patients, it increases the risk of ovarian hyperstimulation syndrome (OHSS) due to its longer half-life compared to the naturally secreted Luteinizing Hormone (LH) as well as increased synthesis and secretion of vasoactive substances. Gonadotropin releasing hormone agonist (GnRHa) triggering, as an alternative to hCG triggering for final oocyte maturation in antagonist protocols, enables substantial decrease of this complication in high responders. However, the main disadvantage of using GnRHa for induction of oocyte maturation is significantly lower pregnancy rates compared with hCG triggering. The primary hypothesis is luteal insufficiency due to increased luteolysis. In order to preserve a high pregnancy rates after GnRHa triggering, several approaches for luteal-phase rescue have been investigated, including low-dose hCG boluses, intensive P and E2 supplementation, and a ''freeze-all'' approach with frozen-thawed embryo transfers at subsequent cycles. Several previous case reports have demonstrated that inadvertent administration of GnRH agonists during the luteal phase doesn't harm pregnancies achieved through IVF and moreover might even support implantation.

The mechanism by which GnRH agonist improve implantation rates is unknown. Several hypotheses were suggested including promoting corpus luteum maintenance by secretion of LH from pituitary gonadotropin cells, a direct effect on the endometrium and the embryo through GnRH receptors and regulatory effect on hCG secretion by the placenta at the preimplantation phase. In 2004, Tesarik et al, conducted a prospective randomized trial including 276 oocyte recipients. Oocytes from each individual donor were divided to two recipients, one of whom received a single dose of a GnRH agonist (0.1 mg triptorelin) 3 days after embryo transfer and the other received placebo at the same time. Of note, the endometrium was prepared by oral estradiol valerate treatment following by vaginal progesterone (Utrogestan) as widely accepted. The results demonstrated significantly higher implantation and live birth rate in the group treated with GnRH agonist compared to the control group with significantly higher twin pregnancy rates while no difference in miscarriage and abortion rates was observed between the two study groups. The authors concluded that GnRH agonist administration at the time of implantation has a positive effect on embryo developmental potential. It's important to note that this study evaluated the effect of a single dose of GnRH agonist in addition to a conventional luteal support in a population of oocyte recipients that are not at risk for OHSS and tend to have higher implantation and pregnancy rates also without GnRH agonist supplementation. A study by Pirard et al. was the first to evaluate the administration of GnRH agonist alone for luteal support compared to compared to the standard treatment with vaginal progesterone. The study group included 35 patients who were treated with antagonist protocol. Intranasal GnRH agonist (Buserilin) was given for final oocyte maturation and luteal support was achieved by administration of intranasal GnRH agonist for up to 16 days after the oocytes retrieval. The control group included 18 women treated with a long GnRH protocol for pituitary suppression. Final oocytes maturation was achieved by administration of 10000 units of hCG and vaginal progesterone was used for luteal support. Implantation and pregnancy rates were higher among the study group compared to the control group however, no statistical significance was achieved. Progesterone levels on day 5 were significantly lower while LH levels were significantly higher during all the luteal phase in the study group compared to the control group. The authors concluded that intranasal administration of Buserelin is as effective as standard progesterone treatment for providing luteal phase support in IVF/ICSI antagonist protocols. To our knowledge, the only study, so far that evaluated the efficacy of GnRH agonist treatment for luteal support in high responder patients with increased risk for OHSS was conducted by Bar-Hava et al. It included 46 women at risk for OHSS that were treated with GnRH antagonist protocol for pituitary suppression. The final oocyte maturation was achieved by GnRH agonist (Triptorelin) and a daily intranasal GnRH agonist (Nafarelin 200 micrograms twice daily) was administered for luteal support for two weeks following the oocytes retrieval. 52% clinical pregnancy rates were obtained while no cases od OHSS or other substantial adverse effects were observed.

The main disadvantage of the study is the lack of a comparison to a control group. To the best of our knowledge, no study so far compared administration of GnRH agonist at the same protocol described by Bar-Hava et al. to intensive estrogen and progesterone treatment for luteal support among women treated with GnRH antagonist protocol and GnRH agonist triggering for final oocytes maturation. A randomized controlled trial in an infertility population at increased risk for OHSS, will enable us to evaluate the efficacy of GnRH agonist treatment compared to standard treatment for luteal support and to determine the best treatment approach in the high responder population undergoing a fresh embryo transfer new approach undergoing a fresh embryo transfer following GnRHa triggering.

The aim of the current study isto compare the efficacy of GnRH agonist versus estrogen and progesterone supplementation for luteal support in high responders undergoing fresh embryo transfer following GnRHa triggering.

ELIGIBILITY:
Inclusion Criteria:

* High responder patients, defined as either reaching a serum estradiol levels of ≥ 3500 pg/ml on the day of trigger or having ≥ 15 oocytes retrieved.
* Increased risk for OHSS (PCOS, previous history of OHSS, high antral follicle count (AFC) etc.).

Exclusion Criteria:

* Repeated implantation failure (3 or more previous failed embryo transfer cycles while transferring good quality embryos).
* Oocyte donation, fertility preservation or Freeze all (freezing all the embryos) cycles.
* Moderate to severe endometriosis
* An evidence of hydrosalpinx

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-29 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 3 weeks after positive serum bHCG results
  an ultrasound visualization of one or more gestational sacs
Clinical pregnancy rate with fetal heart beat | 3 weeks after positive serum bHCG results
  clinical pregnancy with a demonstration of fetal heart by ultrasound visualization

SECONDARY OUTCOMES:
Miscarriage rate | from the demonstration of a clinical pregnancy (3 weeks after positive serum bHCG results) up to 22 weeks
  spontaneous loss of a clinical pregnancy before 22 completed weeks of gestational age
Ovarian hyperstimulation syndrome (OHSS) rate | up to 12 days post embryo transfer
  An exaggerated systemic response to ovarian stimulation characterized by a wide spectrum of clinical and laboratory manifestations. It may be classified as mild, moderate or severe according to the degree of abdominal distention, ovarian enlargement and respiratory, hemodynamic and metabolic complications.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Youngster, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gomez R, Soares SR, Busso C, Garcia-Velasco JA, Simon C, Pellicer A. Physiology and pathology of ovarian hyperstimulation syndrome. Semin Reprod Med. 2010 Nov;28(6):448-57. doi: 10.1055/s-0030-1265670. Epub 2010 Nov 16. PMID 21082502
- [Background] Damewood MD, Shen W, Zacur HA, Schlaff WD, Rock JA, Wallach EE. Disappearance of exogenously administered human chorionic gonadotropin. Fertil Steril. 1989 Sep;52(3):398-400. doi: 10.1016/s0015-0282(16)60906-8. PMID 2776893
- [Background] Leth-Moller K, Hammer Jagd S, Humaidan P. The Luteal Phase after GnRHa Trigger-Understanding An Enigma. Int J Fertil Steril. 2014 Oct;8(3):227-34. Epub 2014 Nov 1. PMID 25379149
- [Background] Youssef MA, Van der Veen F, Al-Inany HG, Mochtar MH, Griesinger G, Nagi Mohesen M, Aboulfoutouh I, van Wely M. Gonadotropin-releasing hormone agonist versus HCG for oocyte triggering in antagonist-assisted reproductive technology. Cochrane Database Syst Rev. 2014 Oct 31;2014(10):CD008046. doi: 10.1002/14651858.CD008046.pub4. PMID 25358904
- [Background] Atkinson P, Koch J, Ledger WL. GnRH agonist trigger and a freeze-all strategy to prevent ovarian hyperstimulation syndrome: a retrospective study of OHSS risk and pregnancy rates. Aust N Z J Obstet Gynaecol. 2014 Dec;54(6):581-5. doi: 10.1111/ajo.12277. PMID 25476811
- [Background] van der Linden M, Buckingham K, Farquhar C, Kremer JA, Metwally M. Luteal phase support for assisted reproduction cycles. Cochrane Database Syst Rev. 2015 Jul 7;2015(7):CD009154. doi: 10.1002/14651858.CD009154.pub3. PMID 26148507
- [Background] Golan A, Ron-el R, Herman A, Weinraub Z, Soffer Y, Caspi E. Fetal outcome following inadvertant administration of long-acting DTRP6 GnRH microcapsules during pregnancy: a case report. Hum Reprod. 1990 Jan;5(1):123-4. doi: 10.1093/oxfordjournals.humrep.a137031. PMID 2139040
- [Background] Isherwood PJ, Ibrahim ZH, Matson PL, Morroll DR, Burslem RW, Lieberman BA. Endocrine changes in women conceiving during treatment with an LHRH agonist. Hum Reprod. 1990 May;5(4):409-12. doi: 10.1093/oxfordjournals.humrep.a137112. PMID 2113928
- [Background] Jackson AE, Curtis P, Amso N, Shaw RW. Exposure to LHRH agonists in early pregnancy following the commencement of mid-luteal buserelin for IVF stimulation. Hum Reprod. 1992 Oct;7(9):1222-4. doi: 10.1093/oxfordjournals.humrep.a137830. PMID 1479001
- [Background] Elefant E, Biour B, Blumberg-Tick J, Roux C, Thomas F. Administration of a gonadotropin-releasing hormone agonist during pregnancy: follow-up of 28 pregnancies exposed to triptoreline. Fertil Steril. 1995 May;63(5):1111-3. doi: 10.1016/s0015-0282(16)57557-8. PMID 7720926
- [Background] Balasch J, Martinez F, Jove I, Cabre L, Coroleu B, Barri PN, Vanrell JA. Inadvertent gonadotrophin-releasing hormone agonist (GnRHa) administration in the luteal phase may improve fecundity in in-vitro fertilization patients. Hum Reprod. 1993 Jul;8(7):1148-51. doi: 10.1093/oxfordjournals.humrep.a138210. PMID 8408503
- [Background] Wilshire GB, Emmi AM, Gagliardi CC, Weiss G. Gonadotropin-releasing hormone agonist administration in early human pregnancy is associated with normal outcomes. Fertil Steril. 1993 Dec;60(6):980-3. doi: 10.1016/s0015-0282(16)56396-1. PMID 8243703
- [Background] Weissman A, Shoham Z. Favourable pregnancy outcome after administration of a long-acting gonadotrophin-releasing hormone agonist in the mid-luteal phase. Hum Reprod. 1993 Mar;8(3):496-7. doi: 10.1093/oxfordjournals.humrep.a138079. PMID 7682565
- [Background] Young DC, Snabes MC, Poindexter AN 3rd. GnRH agonist exposure during the first trimester of pregnancy. Obstet Gynecol. 1993 Apr;81(4):587-9. PMID 8459972
- [Background] Gartner B, Moreno C, Marinaro A, Remohi J, Simon C, Pellicer A. Accidental exposure to daily long-acting gonadotrophin-releasing hormone analogue administration and pregnancy in an in-vitro fertilization cycle. Hum Reprod. 1997 Nov;12(11):2557-9. doi: 10.1093/humrep/12.11.2557. PMID 9436706
- [Background] Tesarik J, Hazout A, Mendoza C. Enhancement of embryo developmental potential by a single administration of GnRH agonist at the time of implantation. Hum Reprod. 2004 May;19(5):1176-80. doi: 10.1093/humrep/deh235. Epub 2004 Apr 7. PMID 15070873
- [Background] Tesarik J, Hazout A, Mendoza-Tesarik R, Mendoza N, Mendoza C. Beneficial effect of luteal-phase GnRH agonist administration on embryo implantation after ICSI in both GnRH agonist- and antagonist-treated ovarian stimulation cycles. Hum Reprod. 2006 Oct;21(10):2572-9. doi: 10.1093/humrep/del173. Epub 2006 Aug 22. PMID 16926261
- [Background] Pirard C, Loumaye E, Laurent P, Wyns C. Contribution to More Patient-Friendly ART Treatment: Efficacy of Continuous Low-Dose GnRH Agonist as the Only Luteal Support-Results of a Prospective, Randomized, Comparative Study. Int J Endocrinol. 2015;2015:727569. doi: 10.1155/2015/727569. Epub 2015 Apr 5. PMID 25945092
- [Background] Bar-Hava I, Mizrachi Y, Karfunkel-Doron D, Omer Y, Sheena L, Carmon N, Ben-David G. Intranasal gonadotropin-releasing hormone agonist (GnRHa) for luteal-phase support following GnRHa triggering, a novel approach to avoid ovarian hyperstimulation syndrome in high responders. Fertil Steril. 2016 Aug;106(2):330-3. doi: 10.1016/j.fertnstert.2016.04.004. Epub 2016 Apr 22. PMID 27114332